CLINICAL TRIAL: NCT03155620
Title: NCI-COG Pediatric MATCH (Molecular Analysis for Therapy Choice) Screening Protocol
Brief Title: Targeted Therapy Directed by Genetic Testing in Treating Pediatric Patients With Relapsed or Refractory Advanced Solid Tumors, Non-Hodgkin Lymphomas, or Histiocytic Disorders (The Pediatric MATCH Screening Trial)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: NCI-2017-01251; NCI-2017-01251 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); APEC1621SC (Other: Children's Oncology Group); APEC1621SC (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2017-05-15; First posted 2017-05-16 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Advanced Malignant Solid Neoplasm; Ann Arbor Stage III Non-Hodgkin Lymphoma; Ann Arbor Stage IV Non-Hodgkin Lymphoma; Histiocytic Sarcoma; Juvenile Xanthogranuloma; Langerhans Cell Histiocytosis; Malignant Glioma; Recurrent Childhood Rhabdomyosarcoma; Recurrent Ependymoma; Recurrent Ewing Sarcoma; Recurrent Glioma; Recurrent Hepatoblastoma; Recurrent Langerhans Cell Histiocytosis; Recurrent Malignant Germ Cell Tumor; Recurrent Malignant Solid Neoplasm; Recurrent Medulloblastoma; Recurrent Neuroblastoma; Recurrent Non-Hodgkin Lymphoma; Recurrent Osteosarcoma; Recurrent Peripheral Primitive Neuroectodermal Tumor; Recurrent Primary Central Nervous System Neoplasm; Recurrent Rhabdoid Tumor; Recurrent Soft Tissue Sarcoma; Refractory Ewing Sarcoma; Refractory Glioma; Refractory Hepatoblastoma; Refractory Langerhans Cell Histiocytosis; Refractory Malignant Germ Cell Tumor; Refractory Malignant Solid Neoplasm; Refractory Medulloblastoma; Refractory Neuroblastoma; Refractory Non-Hodgkin Lymphoma; Refractory Osteosarcoma; Refractory Peripheral Primitive Neuroectodermal Tumor; Refractory Primary Central Nervous System Neoplasm; Refractory Rhabdoid Tumor; Refractory Rhabdomyosarcoma; Rhabdoid Tumor; Stage III Osteosarcoma AJCC v7; Stage III Soft Tissue Sarcoma AJCC v7; Stage IV Osteosarcoma AJCC v7; Stage IV Soft Tissue Sarcoma AJCC v7; Stage IVA Osteosarcoma AJCC v7; Stage IVB Osteosarcoma AJCC v7; Wilms Tumor
MeSH Terms: conditions — Histiocytic Sarcoma; Xanthogranuloma, Juvenile; Histiocytosis, Langerhans-Cell; Glioma; Ependymoma; Sarcoma, Ewing; Hepatoblastoma; Medulloblastoma; Neuroblastoma; Lymphoma, Non-Hodgkin; Osteosarcoma; Neuroectodermal Tumors, Primitive, Peripheral; Central Nervous System Neoplasms; Rhabdoid Tumor; Sarcoma; Rhabdomyosarcoma; Wilms Tumor | interventions — Biopsy; Specimen Handling; ensartinib; erdafitinib; ivosidenib; larotrectinib; Magnetic Resonance Spectroscopy; olaparib; palbociclib; Nuclear Medicine Department, Hospital; LY3023414; selpercatinib; tazemetostat; tipifarnib; ulixertinib; Vemurafenib; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Subprotocol A (NTRK1, NTRK2, or NTRK3 gene fusion) (Experimental): Patients with a NTRK1, NTRK2, or NTRK3 gene fusion receive larotrectinib sulfate PO or via nasogastric- or gastric-tube BID on days 1-28. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis; Drug: Larotrectinib Sulfate; Procedure: Mutation Carrier Screening; Other: Pharmacological Study
- Subprotocol B (FGFR1, FGFR2, FGFR3, or FGFR4 gene mutation) (Experimental): Patients with a FGFR1, FGFR2, FGFR3, or FGFR4 gene mutation receive erdafitinib PO QD on days 1-28 of each cycle. Treatment repeats every 28 days for up to 26 cycles (2 years) in the absence of disease progression or unacceptable toxicity. Patients undergo an x-ray, CT scan, MRI, radionuclide imaging, and/or bone scan, as well as a bone marrow aspiration and/or biopsy during screening and on study. Patients also undergo blood sample collection on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Erdafitinib; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Procedure: Mutation Carrier Screening; Other: Pharmacological Study; Procedure: Radionuclide Imaging; Procedure: X-Ray Imaging
- Subprotocol C (EZH2, SMARCB1, or SMARCA4 gene mutation) (Experimental): Patients with an EZH2, SMARCB1, or SMARCA4 gene mutation receive tazemetostat PO BID on days 1-28. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis; Procedure: Mutation Carrier Screening; Other: Pharmacological Study; Drug: Tazemetostat
- Subprotocol D (TSC1, TSC2, or PI3K/mTOR gene mutation) (Experimental): Patients with a TSC1, TSC2, or PI3K/mTOR gene mutations receive PI3K/mTOR inhibitor LY3023414 PO BID on days 1-28. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis; Procedure: Mutation Carrier Screening; Other: Pharmacological Study; Drug: Samotolisib
- Subprotocol E (activating MAPK pathway gene mutation) (Experimental): Patients with an activating MAPK pathway gene mutation receive selumetinib sulfate PO BID on days 1-28. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis; Procedure: Mutation Carrier Screening; Other: Pharmacological Study; Drug: Selumetinib Sulfate
- Subprotocol F (ALK or ROS1 gene alteration) (Experimental): Patients with an ALK or ROS1 gene alteration receive ensartinib PO BID on days 1-28. Cycles repeat every 28 days for 2 years (up to 26 cycles) in the absence of disease progression or unacceptable toxicity. Patients undergo an x-ray, CT scan, MRI, PET scan, radionuclide imaging, and/or bone scan, as well as a bone marrow aspiration and/or biopsy during screening and on study. Patients also undergo blood sample collection on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Ensartinib; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Procedure: Mutation Carrier Screening; Other: Pharmacological Study; Procedure: Positron Emission Tomography; Procedure: Radionuclide Imaging; Procedure: X-Ray Imaging
- Subprotocol G (BRAF V600 gene mutation) (Experimental): Patients with a BRAF V600 gene mutation receive vemurafenib PO BID on days 1-28. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis; Procedure: Mutation Carrier Screening; Other: Pharmacological Study; Drug: Vemurafenib
- Subprotocol H (ATM, BRCA1, BRCA2, RAD51C, RAD51D mutations) (Experimental): Patients deleterious ATM, BRCA1, BRCA2, RAD51C, or RAD51D gene mutations receive olaparib PO BID on days 1-28. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis; Procedure: Mutation Carrier Screening; Drug: Olaparib; Other: Pharmacological Study
- Subprotocol I (Rb positive, alterations in cell cycle genes) (Experimental): Patients with Rb positive advanced solid tumors, non-Hodgkin lymphoma, or histiocytic disorders with activating alterations in cell cycle genes receive palbociclib PO QD on days 1-21. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis; Procedure: Mutation Carrier Screening; Drug: Palbociclib; Other: Pharmacological Study
- Subprotocol J (MAPK pathway mutations) (Experimental): Patients with MAPK pathway mutations receive ulixertinib PO BID. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis; Procedure: Mutation Carrier Screening; Other: Pharmacological Study; Drug: Ulixertinib
- Subprotocol K (IDH1 gene mutation) (Experimental): Patients with IDH1 gene mutations receive ivosidenib PO QD. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Ivosidenib; Other: Laboratory Biomarker Analysis; Procedure: Mutation Carrier Screening; Other: Pharmacological Study
- Subprotocol M (HRAS gene alterations) (Experimental): Patients receive tipifarnib PO or via nasogastric or gastric tube BID on days 1-7 and 15-21. Treatment repeats every 28 days for up to 26 cycles (2 years) in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis; Procedure: Mutation Carrier Screening; Other: Pharmacological Study; Drug: Tipifarnib
- Subprotocol N (activating RET mutations) (Experimental): Patients with activating RET gene alterations receive selpercatinib PO BID on days 1-28. Treatment repeats every 28 days for up to 26 cycles (2 years) in the absence of disease progression or unacceptable toxicity. Patients may also undergo PET, CT, MRI, PET/CT, PET/MRI, and/or CT/MRI, scintigraphy, and x-ray imaging throughout the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Procedure: Mutation Carrier Screening; Other: Pharmacological Study; Procedure: Positron Emission Tomography; Procedure: Radionuclide Imaging; Drug: Selpercatinib; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration and Biopsy — Undergo a bone marrow and/or biopsy
  Arms: Subprotocol B (FGFR1, FGFR2, FGFR3, or FGFR4 gene mutation); Subprotocol F (ALK or ROS1 gene alteration)
Procedure: Bone Scan — Undergo a bone scan
  Other Names: Bone Scintigraphy
  Arms: Subprotocol B (FGFR1, FGFR2, FGFR3, or FGFR4 gene mutation); Subprotocol F (ALK or ROS1 gene alteration)
Procedure: Computed Tomography — Undergo CT, PET/Ct, and/or CT/MRI
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
  Arms: Subprotocol B (FGFR1, FGFR2, FGFR3, or FGFR4 gene mutation); Subprotocol F (ALK or ROS1 gene alteration); Subprotocol N (activating RET mutations)
Drug: Ensartinib — Given PO
  Other Names: X 396; X-396; X396
  Arms: Subprotocol F (ALK or ROS1 gene alteration)
Drug: Erdafitinib — Given PO
  Other Names: Balversa; JNJ 42756493; JNJ-42756493; JNJ42756493
  Arms: Subprotocol B (FGFR1, FGFR2, FGFR3, or FGFR4 gene mutation)
Drug: Ivosidenib — Given PO
  Other Names: AG 120; AG-120; AG120; Tibsovo
  Arms: Subprotocol K (IDH1 gene mutation)
Other: Laboratory Biomarker Analysis — Undergo molecular analysis
Drug: Larotrectinib Sulfate — Given PO or via nasogastric- or gastric-tube
  Other Names: ARRY 470 Sulfate; LOXO 101 Sulfate; LOXO-101 Sulfate; Vitrakvi
  Arms: Subprotocol A (NTRK1, NTRK2, or NTRK3 gene fusion)
Procedure: Magnetic Resonance Imaging — Undergo MRI, PET/MRI, and/or CT/MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
  Arms: Subprotocol B (FGFR1, FGFR2, FGFR3, or FGFR4 gene mutation); Subprotocol F (ALK or ROS1 gene alteration); Subprotocol N (activating RET mutations)
Procedure: Mutation Carrier Screening — Undergo tumor tissue mutation screening
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU 0059436; KU-0059436; KU0059436; Lynparza; Olanib; Olaparix; PARP Inhibitor AZD2281
  Arms: Subprotocol H (ATM, BRCA1, BRCA2, RAD51C, RAD51D mutations)
Drug: Palbociclib — Given PO
  Other Names: 6-Acetyl-8-cyclopentyl-5-methyl-2-((5-(piperazin-1-yl)pyridin-2-yl)amino)-8h-pyrido(2,3-d)pyrimidin-7-one; Ibrance; PD 0332991; PD 332991; PD 991; PD-0332991; PD0332991
  Arms: Subprotocol I (Rb positive, alterations in cell cycle genes)
Other: Pharmacological Study — Correlative studies
Procedure: Positron Emission Tomography — Undergo PET, PET/CT, and/or PET/MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
  Arms: Subprotocol F (ALK or ROS1 gene alteration); Subprotocol N (activating RET mutations)
Procedure: Radionuclide Imaging — Undergo radionuclide imaging
  Other Names: NM; Nuclear Medicine; nuclear medicine scan; radioimaging; Radionuclide Scanning; Scan; Scintigraphy
  Arms: Subprotocol B (FGFR1, FGFR2, FGFR3, or FGFR4 gene mutation); Subprotocol F (ALK or ROS1 gene alteration); Subprotocol N (activating RET mutations)
Drug: Samotolisib — Given PO
  Other Names: 2H-Imidazo(4,5-C)quinolin-2-one, 1,3-Dihydro-8-(5-(1-hydroxy-1-methylethyl)-3-pyridinyl)-1-((2S)-2-methoxypropyl)-3-methyl-; LY 3023414; LY-3023414; LY3023414; WHO 10889
  Arms: Subprotocol D (TSC1, TSC2, or PI3K/mTOR gene mutation)
Drug: Selpercatinib — Given PO
  Other Names: LOXO 292; LOXO-292; LOXO292; RET Kinase Inhibitor LOXO-292; Retevmo; Retsevmo; WHO 10967
  Arms: Subprotocol N (activating RET mutations)
Drug: Selumetinib Sulfate — Given PO
  Other Names: AZD-6244 Hydrogen Sulfate; AZD6244 Hydrogen Sulfate; AZD6244 Hydrogen Sulphate; Koselugo; Selumetinib Sulphate
  Arms: Subprotocol E (activating MAPK pathway gene mutation)
Drug: Tazemetostat — Given PO
  Other Names: E 7438; E-7438; E7438; EPZ 6438; EPZ-6438; EPZ6438
  Arms: Subprotocol C (EZH2, SMARCB1, or SMARCA4 gene mutation)
Drug: Tipifarnib — Given PO or via nasogastric or gastric tube
  Other Names: R115777; Zarnestra
  Arms: Subprotocol M (HRAS gene alterations)
Drug: Ulixertinib — Receive PO
  Other Names: BVD-523; VRT752271
  Arms: Subprotocol J (MAPK pathway mutations)
Drug: Vemurafenib — Given PO
  Other Names: BRAF (V600E) kinase inhibitor RO5185426; BRAF(V600E) Kinase Inhibitor RO5185426; PLX 4032; PLX-4032; PLX4032; RG 7204; RG-7204; RG7204; RO 5185426; RO-5185426; Zelboraf
  Arms: Subprotocol G (BRAF V600 gene mutation)
Procedure: X-Ray Imaging — Undergo an x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray
  Arms: Subprotocol B (FGFR1, FGFR2, FGFR3, or FGFR4 gene mutation); Subprotocol F (ALK or ROS1 gene alteration); Subprotocol N (activating RET mutations)

SUMMARY:
This phase II Pediatric MATCH screening and multi-sub-trial studies how well treatment that is directed by genetic testing works in pediatric patients with solid tumors, non-Hodgkin lymphomas, or histiocytic disorders that have progressed following at least one line of standard systemic therapy and/or for which no standard treatment exists that has been shown to prolong survival. Genetic tests look at the unique genetic material (genes) of patients' tumor cells. Patients with genetic changes or abnormalities (mutations) may benefit more from treatment which targets their tumor's particular genetic mutation, and may help doctors plan better treatment for patients with solid tumors or non-Hodgkin lymphomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To utilize clinical and biological data to screen for eligibility to phase 2 pathway-targeting specific subprotocols of pathway-targeting agents in pediatric patients with advanced solid tumors, non-Hodgkin lymphomas, and histiocytic disorders.

II. To determine the proportion of pediatric patients whose advanced tumors have pathway alterations that can be targeted by select anti-cancer drugs. (Completed as of Amendment #4. Patients enrolled on or after Amendment 4 will not be included in this analysis as screening of unselected patients will no longer be conducted.)

SECONDARY OBJECTIVE:

I. To obtain preliminary information on the response rate to targeted therapy in patients whose tumors lack actionable alterations as defined for the molecular analysis for therapy choice (MATCH) study, for selected agents for which efficacy is observed in the primary matched cohort.

EXPLORATORY OBJECTIVES:

I. To increase knowledge of the genomic landscape of advanced pediatric solid tumors, non-Hodgkin lymphomas, and histiocytic disorders.

II. To describe the genomic changes that occur in advanced pediatric cancers between the time of initial diagnosis and relapse, in cases for which paired tumor specimens are available.

III. To explore approaches to diagnosing and profiling genomics of advanced pediatric cancers through evaluation of circulating tumor deoxyribonucleic acid (DNA).

IV. To determine the frequency and spectrum of germline cancer susceptibility mutations in children with relapsed solid tumors and non-Hodgkin lymphomas and assess the feasibility of return of those results in the National Clinical Trial Network (NCTN) group setting.

OUTLINE:

STEP 1 (SCREENING): Patients undergo biopsy along with tumor mutational screening of the biopsy material for specific, pre-defined mutations, amplifications, or translocations of interest via tumor sequencing and immunohistochemistry. Patients also undergo collection of blood samples for research purposes.

STEP 2 (TREATMENT): Patients with a mutation targeted by one or more of the investigational drugs used in this study or those without mutations are assigned to 1 of 13 treatment subprotocols.

APEC1621A: Patients with a NTRK1, NTRK2, or NTRK3 gene fusion receive larotrectinib sulfate orally (PO) or via nasogastric- or gastric-tube twice daily (BID) on days 1-28. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.

APEC1621B: Patients with a FGFR1, FGFR2, FGFR3, or FGFR4 gene mutation receive erdafitinib PO once daily (QD) on days 1-28 of each cycle. Treatment repeats every 28 days for up to 26 cycles (2 years) in the absence of disease progression or unacceptable toxicity. Patients undergo an x-ray, computed tomography (CT scan), magnetic resonance imaging (MRI), radionuclide imaging, and/or bone scan, as well as a bone marrow aspiration and/or biopsy during screening and on study. Patients also undergo blood sample collection on study.

APEC1621C: Patients with an EZH2, SMARCB1, or SMARCA4 gene mutation receive tazemetostat PO BID on days 1-28. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.

APEC1621D: Patients with a TSC1, TSC2, or PI3K/mTOR gene mutations receive PI3K/mTOR inhibitor LY3023414 PO BID on days 1-28. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.

APEC1621E: Patients with an activating MAPK pathway gene mutation receive selumetinib sulfate PO BID on days 1-28. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.

APEC1621F: Patients with an ALK or ROS1 gene alteration receive ensartinib (ALK Inhibitor X-396) PO BID on days 1-28. Cycles repeat every 28 days for 2 years (up to 26 cycles) in the absence of disease progression or unacceptable toxicity. Patients undergo an x-ray, CT scan, MRI, PET scan, radionuclide imaging, and/or bone scan, as well as a bone marrow aspiration and/or biopsy during screening and on study. Patients also undergo blood sample collection on study.

APEC1621G: Patients with a BRAF V600 gene mutation receive vemurafenib PO BID on days 1-28. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.

APEC1621H: Patients with deleterious ATM, BRCA1, BRCA2, RAD51C, or RAD51D gene mutations receive olaparib PO BID on days 1-28. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.

APEC1621I: Patients with Rb positive advanced solid tumors, non-Hodgkin lymphoma, or histiocytic disorders with activating alterations in cell cycle genes receive palbociclib PO QD on days 1-21. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

APEC1621J: Patients with MAPK Pathway Mutations receive ulixertinib PO BID. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

APEC1621K: Patients with IDH1 gene mutations receive ivosidenib PO QD. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

APEC1621M: Patients with HRAS gene alterations receive tipifarnib PO or via nasogastric or gastric tube BID on days 1-7 and 15-21. Treatment repeats every 28 days for up to 26 cycles (2 years) in the absence of disease progression or unacceptable toxicity.

APEC1621N: Patients with activating RET gene alterations receive selpercatinib PO BID on days 1-28. Treatment repeats every 28 days for up to 26 cycles (2 years) in the absence of disease progression or unacceptable toxicity. Patients may also undergo PET, CT, MRI, PET/CT, PET/MRI, and/or CT/MRI, scintigraphy, and x-ray imaging throughout the trial.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* ELIGIBILITY CRITERIA FOR ENROLLMENT ONTO APEC1621SC: Patients must be >= 12 months and =< 21 years of age at the time of study enrollment
* ELIGIBILITY CRITERIA FOR ENROLLMENT ONTO APEC1621SC: Patients with recurrent or refractory solid tumors, including non-Hodgkin lymphomas, histiocytoses (e.g. langerhans cell histiocytosis [LCH], juvenile xanthogranuloma [JXG], histiocytic sarcoma), and central nervous system (CNS) tumors are eligible; patients must have had histologic verification of malignancy at original diagnosis or relapse except in patients with intrinsic brain stem tumors, optic pathway gliomas, or patients with pineal tumors and elevations of cerebrospinal fluid (CSF) or serum tumor markers including alpha-fetoprotein or beta-human chorionic gonadotropin (HCG); in cases where patient enrolls prior to histologic confirmation of recurrent disease, patient is ineligible and should be withdrawn from study if histology fails to confirm recurrence; please note: Patients with Hodgkin lymphoma and plexiform neurofibroma are not eligible
* ELIGIBILITY CRITERIA FOR ENROLLMENT ONTO APEC1621SC: Tumor Testing Requirement: Tumor sample availability requirement for stage 1 of Pediatric MATCH (patients enrolled from start of study in July 2017 through 12/31/21); Patients must have an formalin-fixed paraffin-embedded (FFPE) tumor sample available for MATCH study testing from a biopsy or surgery that was performed at any point after initial tumor recurrence/progression, or be planned to have a procedure to obtain such a sample that is considered to be of potential benefit by the treating clinicians; a tumor sample from a clinically performed diagnostic (pre-treatment) biopsy will be acceptable for enrollment onto Pediatric MATCH only for children with high-grade gliomas of the brainstem (diffuse intrinsic pontine gliomas) or thalamus

  * Please note: Samples that have been decalcified using standardly utilized acid-based decalcification methods are not generally suitable for MATCH study testing; the nucleic acids will have been degraded in the decalcification process
* ELIGIBILITY CRITERIA FOR ENROLLMENT ONTO APEC1621SC: Tumor molecular profiling report availability requirement for Stage 2 of Pediatric MATCH (patients enrolled starting 2022): In stage 2 of the study, no tumor samples will be submitted for centralized clinical tumor profiling; instead, a tumor molecular profiling report from a College of American Pathologists (CAP)/ Clinical Laboratory Improvements Amendments (CLIA)-approved testing laboratory must be submitted for review by the Molecular Review Committee (MRC)

  * This molecular profiling must have been performed on a tumor sample that was obtained at any point after initial tumor recurrence/progression and must be accompanied by a pathology report for the same tumor specimen; a molecular profiling report for a diagnostic (pre-treatment) tumor sample will be acceptable for enrollment onto Pediatric MATCH only for children with high-grade gliomas of the brainstem (diffuse intrinsic pontine gliomas) or thalamus. In the event that molecular profiling reports are available from multiple timepoints, the most recent report should be prioritized for study submission
* ELIGIBILITY CRITERIA FOR ENROLLMENT ONTO APEC1621SC: Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age); note: neurologic deficits in patients with CNS tumors must have been stable for at least 7 days prior to study enrollment; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* ELIGIBILITY CRITERIA FOR ENROLLMENT ONTO APEC1621SC: Patients must have radiographically measurable disease; measurable disease based on imaging obtained less than or equal to 56 days prior to enrollment; patients with neuroblastoma who do not have measurable disease but have metaiodobenzylguanidine (MIBG) positive (+) evaluable disease are eligible; measurable disease in patients with CNS involvement is defined as any lesion that is at minimum 10 mm in one dimension on standard magnetic resonance imaging (MRI) or computed tomography (CT)

  * Note: The following do not qualify as measurable disease:

    * Malignant fluid collections (e.g., ascites, pleural effusions)
    * Bone marrow infiltration except that detected by MIBG scan for neuroblastoma
    * Lesions only detected by nuclear medicine studies (e.g., bone, gallium or positron emission tomography [PET] scans) except as noted for neuroblastoma
    * Elevated tumor markers in plasma or CSF
    * Previously radiated lesions that have not demonstrated clear progression post radiation
    * Leptomeningeal lesions that do not meet the measurement requirements for Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* GENERAL INCLUSION CRITERIA FOR SUBPROTOCOLS: NOTE: patient does not need to meet all subprotocol criteria at time of enrollment onto the APEC1621SC screening protocol, but will need to meet all criteria prior to enrollment on any assigned treatment subprotocol. Patients must be enrolled onto a subprotocol within 2 weeks (14 days) of treatment assignment
* GENERAL INCLUSION CRITERIA FOR SUBPROTOCOLS: Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age); Note: neurologic deficits in patients with CNS tumors must have been stable for at least 7 days prior to study enrollment; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* GENERAL INCLUSION CRITERIA FOR SUBPROTOCOLS: At the time of treatment with subprotocol specified therapy, the patients must have radiographically measurable disease; patients with neuroblastoma who do not have measurable disease but have MIBG+ evaluable are eligible; measurable disease in patients with CNS involvement is defined as any lesion that is at minimum 10 mm in one dimension on standard MRI or CT

  * Note: The following do not qualify as measurable disease:

    * Malignant fluid collections (e.g., ascites, pleural effusions)
    * Bone marrow infiltration except that detected by MIBG scan for neuroblastoma
    * Lesions only detected by nuclear medicine studies (e.g., bone, gallium or positron emission tomography [PET] scans) except as noted for neuroblastoma
    * Elevated tumor markers in plasma or CSF
    * Previously radiated lesions that have not demonstrated clear progression post radiation
    * Leptomeningeal lesions that do not meet the measurement requirements for RECIST 1.1
* GENERAL INCLUSION CRITERIA FOR SUBPROTOCOLS: At the time of enrollment onto a subprotocol, the following general criteria for initiation of therapy will be required:

  * Patients must have fully recovered from the acute toxic effects of all prior anticancer therapy and must meet the following minimum duration from prior anticancer directed therapy prior to enrollment to the subprotocol; if after the required timeframe, the numerical eligibility criteria are met, e.g. blood count criteria, the patient is considered to have recovered adequately

    * Cytotoxic chemotherapy or other anticancer agents known to be myelosuppressive: for agents not listed, the duration of this interval must be discussed with the study chair and the study-assigned research coordinator prior to enrollment >= 21 days after the last dose of cytotoxic or myelosuppressive chemotherapy (42 days if prior nitrosourea)
    * Anticancer agents not known to be myelosuppressive (e.g. not associated with reduced platelet or absolute neutrophil counts [ANC]): >= 7 days after the last dose of agent; for agents not listed, the duration of this interval must be discussed with the study chair and the study-assigned research coordinator prior to enrollment
    * Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1
    * Corticosteroids: If used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
    * Hematopoietic growth factors: >= 14 days after the last dose of a long-acting growth factor (e.g. Neulasta) or 7 days for short-acting growth factor; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair and the study-assigned research coordinator
    * Interleukins, interferons and cytokines (other than hematopoietic growth factors): >= 21 days after the completion of interleukins, interferon or cytokines (other than hematopoietic growth factors)
    * Stem cell infusions (with or without total-body irradiation [TBI]):

      * Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including donor lymphocyte infusion (DLI) or boost infusion: >= 84 days after infusion and no evidence of graft versus host disease (GVHD)
      * Autologous stem cell infusion including boost infusion: >= 42 days
    * Cellular therapy: >= 42 days after the completion of any type of cellular therapy (e.g. modified T cells, natural killer (NK) cells, dendritic cells, etc.)
    * X-ray therapy (XRT)/External Beam Irradiation including Protons: >= 14 days after local XRT; >= 150 days after TBI, craniospinal XRT or if radiation to >= 50% of the pelvis; >= 42 days if other substantial bone marrow (BM) radiation; note: radiation may not be delivered to "measurable disease" tumor site(s) being used to follow response to subprotocol treatment
    * Radiopharmaceutical therapy (e.g., radiolabeled antibody, 131I-MIBG): >= 42 days after systemically administered radiopharmaceutical therapy
* GENERAL INCLUSION CRITERIA FOR SUBPROTOCOLS: For patients with solid tumors without known bone marrow involvement:

  * Peripheral absolute neutrophil count (ANC) >= 1000/mm^3
  * Platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* GENERAL INCLUSION CRITERIA FOR SUBPROTOCOLS: Patients with known bone marrow metastatic disease will be eligible for study provided they meet the blood counts (may receive transfusions provided they are not known to be refractory to red cell or platelet transfusions); these patients will not be evaluable for hematologic toxicity
* GENERAL INCLUSION CRITERIA FOR SUBPROTOCOLS: Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 ml/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * Age: 1 to < 2 years; maximum serum creatinine (mg/dL): male 0.6; female 0.6
  * Age: 2 to < 6 years; maximum serum creatinine (mg/dL): male 0.8; female 0.8
  * Age: 6 to < 10 years; maximum serum creatinine (mg/dL): male 1; female 1
  * Age: 10 to < 13 years; maximum serum creatinine (mg/dL): male 1.2; female 1.2
  * Age: 13 to < 16 years; maximum serum creatinine (mg/dL): male 1.5; female 1.4
  * Age: >= 16 years; maximum serum creatinine (mg/dL): male 1.7; female 1.4
* GENERAL INCLUSION CRITERIA FOR SUBPROTOCOLS: Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age
* GENERAL INCLUSION CRITERIA FOR SUBPROTOCOLS: Serum glutamate pyruvate transaminase (SGPT) (alanine transferase [ALT]) =< 135 U/L (for the purpose of this study, the ULN for SGPT is 45 U/L)
* GENERAL INCLUSION CRITERIA FOR SUBPROTOCOLS: Patients must be able to swallow intact capsules/tablets, unless otherwise specified in the subprotocol to which they are assigned
* GENERAL INCLUSION CRITERIA FOR SUBPROTOCOLS: Agent specific limitations on prior therapy will be included with specific treatment subprotocols

Exclusion Criteria:

* GENERAL EXCLUSION CRITERIA FOR SUBPROTOCOLS: Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies, or because there is currently no available information regarding human fetal or teratogenic toxicities; pregnancy tests must be obtained in females who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method
* GENERAL EXCLUSION CRITERIA FOR SUBPROTOCOLS: Concomitant medications

  * Corticosteroids: at the time of consent and enrollment to regimen specific subprotocols, patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment to the subprotocol will not be eligible; if used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
  * Investigational drugs: patients must meet criteria for prior therapy at the time of consent and enrollment to a subprotocol; other investigational agents may not be administered to patients while they are receiving study drug as part of a subprotocol
  * Anticancer agents: patients must meet criteria for prior therapy at the time of consent and enrollment to a subprotocol; other investigational agents may not be administered to patients while they are receiving study drug as part of a subprotocol
  * Anti-GVHD agents post-transplant: patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible
* GENERAL EXCLUSION CRITERIA FOR SUBPROTOCOLS: Patients who have an uncontrolled infection are not eligible
* GENERAL EXCLUSION CRITERIA FOR SUBPROTOCOLS: Patients who have had a prior solid organ transplant are not eligible
* GENERAL EXCLUSION CRITERIA FOR SUBPROTOCOLS: Additional agent specific criteria will be included with specific treatment subprotocols

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1376 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2027-01-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of pediatric patients whose advanced tumors have pathway alterations that can be targeted by select anti-cancer drugs | Up to 2 years from study entry
  Match rate will be calculated as the percent of eligible patients who have an actionable mutation of interest and are matched to at least one of the subprotocols, and confidence intervals will be constructed using the Wilson score interval method. Patients enrolled on or after Amendment 4 will not be included in this analysis as screening of unselected patients will no longer be conducted.

SECONDARY OUTCOMES:
Objective response rate (ORR) to targeted therapy in tumors lacking actionable alterations | Up to 2 years from study entry
  Response rates will be calculated as the percent of evaluable patients who are responders, and confidence intervals will be constructed using the Wilson score interval method.

OTHER OUTCOMES:
Genomic landscape of advanced pediatric solid tumors, non-Hodgkin lymphomas, and histiocytic disorders | Up to 4 years
  A descriptive analysis will be performed and will be summarized with simple summary statistics. This analysis will be descriptive in nature.
Change in genomics in advanced pediatric cancers | Baseline up to 4 years
  A descriptive analysis will be performed and will be summarized with simple summary statistics. This analysis will be descriptive in nature.
Diagnostic and profiling genomics of tumor approach | Up to 4 years
  Will be evaluated through circulating tumor deoxyribonucleic acid (DNA). A descriptive analysis will be performed and will be summarized with simple summary statistics. This analysis will be descriptive in nature.
Frequency of germline cancer susceptibility mutations in children with relapsed solid tumors and non-Hodgkin lymphomas | Up to 4 years
  A descriptive analysis will be performed and will be summarized with simple summary statistics. This analysis will be descriptive in nature. Will assess the feasibility of return of the results in the National Clinical Trial Network (NCTN) group setting.
Spectrum of germline cancer susceptibility mutations in children with relapsed solid tumors and non-Hodgkin lymphomas | Up to 4 years
  A descriptive analysis will be performed and will be summarized with simple summary statistics. This analysis will be descriptive in nature. Will assess the feasibility of return of the results in the NCTN group setting.

CONTACTS AND LOCATIONS:
Overall Officials: Donald W Parsons, Principal Investigator — Children's Oncology Group
Locations (172):
- United States (168):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Perth Children's Hospital, Perth, Western Australia, Australia
- Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec, Canada
- Puerto Rico (2):
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan

REFERENCES:
- [Derived] Scollon S, Plon SE, Joffe S, Biegel JA, Kulkarni S, Miles G, Patton DR, Coffey B, Winter CL, Tsongalis GJ, Routbort MJ, Ramirez NC, Saguilig L, Piao J, Alonzo TA, Berg SL, Fox E, Weigel B, Hawkins DS, Abrams JS, Mooney M, Takebe N, Tricoli JV, Janeway KA, Seibel NL, Parsons DW; NCI-COG Pediatric MATCH Germline Reporting Committee. Germline Cancer Predisposition Results From the National Cancer Institute-Children's Oncology Group Pediatric MATCH Trial. JCO Precis Oncol. 2025 Oct;9:e2500742. doi: 10.1200/PO-25-00742. Epub 2025 Oct 30. PMID 41166674
- [Derived] Parsons DW, Janeway KA, Patton DR, Winter CL, Coffey B, Williams PM, Roy-Chowdhuri S, Tsongalis GJ, Routbort M, Ramirez NC, Saguilig L, Piao J, Alonzo TA, Berg SL, Fox E, Hawkins DS, Abrams JS, Mooney M, Takebe N, Tricoli JV, Seibel NL; NCI-COG Pediatric MATCH Team. Actionable Tumor Alterations and Treatment Protocol Enrollment of Pediatric and Young Adult Patients With Refractory Cancers in the National Cancer Institute-Children's Oncology Group Pediatric MATCH Trial. J Clin Oncol. 2022 Jul 10;40(20):2224-2234. doi: 10.1200/JCO.21.02838. Epub 2022 Mar 30. PMID 35353553
- [Derived] Jain J, Sutton KS, Hong AL. Progress Update in Pediatric Renal Tumors. Curr Oncol Rep. 2021 Feb 16;23(3):33. doi: 10.1007/s11912-021-01016-y. PMID 33591402

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/20/NCT03155620/Prot_SAP_000.pdf